CLINICAL TRIAL: NCT01177371
Title: High-dose Busulfan, High-dose Cyclophosphamide, and Allogeneic Bone Marrow Transplantation for Leukemia, Myelodysplastic Syndromes, Multiple Myeloma and Lymphoma
Brief Title: High-Dose Busulfan and High-Dose Cyclophosphamide Followed By Donor Bone Marrow Transplant in Treating Patients With Leukemia, Myelodysplastic Syndrome, Multiple Myeloma, or Recurrent Hodgkin or Non-Hodgkin Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Lazarus, Hillard, Ireland Cancer Center at University Hospitals Case Medical Center, Case Comprehensive Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CWRU1494T; NCI-2010-01793
Record Dates: First submitted 2010-08-05; First posted 2010-08-09 (Estimated); Last update posted 2010-08-09 (Estimated); Status verified 2010-08

CONDITIONS: Accelerated Phase Chronic Myelogenous Leukemia; Adult Acute Lymphoblastic Leukemia in Remission; Adult Acute Megakaryoblastic Leukemia (M7); Adult Acute Monoblastic Leukemia (M5a); Adult Acute Monocytic Leukemia (M5b); Adult Acute Myeloblastic Leukemia With Maturation (M2); Adult Acute Myeloblastic Leukemia Without Maturation (M1); Adult Acute Myeloid Leukemia in Remission; Adult Acute Myeloid Leukemia With 11q23 (MLL) Abnormalities; Adult Acute Myeloid Leukemia With Del(5q); Adult Acute Myeloid Leukemia With Inv(16)(p13;q22); Adult Acute Myeloid Leukemia With T(15;17)(q22;q12); Adult Acute Myeloid Leukemia With T(16;16)(p13;q22); Adult Acute Myeloid Leukemia With T(8;21)(q22;q22); Adult Acute Myelomonocytic Leukemia (M4); Adult Acute Promyelocytic Leukemia (M3); Adult Erythroleukemia (M6a); Adult Nasal Type Extranodal NK/T-cell Lymphoma; Adult Pure Erythroid Leukemia (M6b); Anaplastic Large Cell Lymphoma; Angioimmunoblastic T-cell Lymphoma; Burkitt Lymphoma; Childhood Acute Erythroleukemia (M6); Childhood Acute Lymphoblastic Leukemia in Remission; Childhood Acute Megakaryocytic Leukemia (M7); Childhood Acute Monoblastic Leukemia (M5a); Childhood Acute Monocytic Leukemia (M5b); Childhood Acute Myeloblastic Leukemia With Maturation (M2); Childhood Acute Myeloblastic Leukemia Without Maturation (M1); Childhood Acute Myeloid Leukemia in Remission; Childhood Acute Myelomonocytic Leukemia (M4); Childhood Acute Promyelocytic Leukemia (M3); Childhood Chronic Myelogenous Leukemia; Childhood Myelodysplastic Syndromes; Chronic Phase Chronic Myelogenous Leukemia; Cutaneous B-cell Non-Hodgkin Lymphoma; De Novo Myelodysplastic Syndromes; Extranodal Marginal Zone B-cell Lymphoma of Mucosa-associated Lymphoid Tissue; Hepatosplenic T-cell Lymphoma; Intraocular Lymphoma; Nodal Marginal Zone B-cell Lymphoma; Peripheral T-Cell Lymphoma; Post-transplant Lymphoproliferative Disorder; Previously Treated Myelodysplastic Syndromes; Recurrent Adult Acute Lymphoblastic Leukemia; Recurrent Adult Acute Myeloid Leukemia; Recurrent Adult Burkitt Lymphoma; Recurrent Adult Diffuse Large Cell Lymphoma; Recurrent Adult Diffuse Mixed Cell Lymphoma; Recurrent Adult Diffuse Small Cleaved Cell Lymphoma; Recurrent Adult Grade III Lymphomatoid Granulomatosis; Recurrent Adult Hodgkin Lymphoma; Recurrent Adult Immunoblastic Large Cell Lymphoma; Recurrent Adult Lymphoblastic Lymphoma; Recurrent Adult Non-Hodgkin Lymphoma; Recurrent Adult T-cell Leukemia/Lymphoma; Recurrent Childhood Acute Lymphoblastic Leukemia; Recurrent Childhood Acute Myeloid Leukemia; Recurrent Cutaneous T-cell Non-Hodgkin Lymphoma; Recurrent Grade 1 Follicular Lymphoma; Recurrent Grade 2 Follicular Lymphoma; Recurrent Grade 3 Follicular Lymphoma; Recurrent Mantle Cell Lymphoma; Recurrent Marginal Zone Lymphoma; Recurrent Mycosis Fungoides/Sezary Syndrome; Recurrent Small Lymphocytic Lymphoma; Refractory Multiple Myeloma; Relapsing Chronic Myelogenous Leukemia; Secondary Myelodysplastic Syndromes; Small Intestine Lymphoma; Splenic Marginal Zone Lymphoma; Testicular Lymphoma; Waldenstrom Macroglobulinemia
MeSH Terms: conditions — Leukemia, Myeloid, Accelerated Phase; Leukemia, Megakaryoblastic, Acute; Leukemia, Monocytic, Acute; Leukemia, Myeloid, Acute; Congenital Abnormalities; Leukemia, Myelomonocytic, Acute; Leukemia, Promyelocytic, Acute; Leukemia, Erythroblastic, Acute; Lymphoma, Extranodal NK-T-Cell; Lymphoma, Large-Cell, Anaplastic; Immunoblastic Lymphadenopathy; Burkitt Lymphoma; Leukemia, Myeloid, Chronic-Phase; Intraocular Lymphoma; Lymphoma, B-Cell, Marginal Zone; Lymphoma, T-Cell, Peripheral; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Hodgkin Disease; Lymphoma, Large-Cell, Immunoblastic; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, T-Cell, Cutaneous; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Mycosis Fungoides; Sezary Syndrome; Leukemia, Lymphocytic, Chronic, B-Cell; Multiple Myeloma; Waldenstrom Macroglobulinemia | interventions — Busulfan; Cyclophosphamide; Transplantation; Methylprednisolone; Methylprednisolone Hemisuccinate; Methylprednisolone Acetate; Methotrexate; merphos; Cyclosporine; Cyclosporins

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm I (Experimental): HIGH-DOSE CHEMOTHERAPY: Patients receive oral busulfan every 6 hours on days -8 to -5 and cyclophosphamide IV over 2 hours on days -4 and -3, or -4 to -2.
  TRANSPLANTATION: Patients undergo allogeneic bone marrow transplant IV over 2-3 hours on day 0.
  GRAFT-VERSUS-HOST DISEASE PROPHYLAXIS: Patients receive cyclosporine IV over 6 hours on day -1, over 10 hours twice daily on days 0-20, and then orally every 12 hours beginning on day 21 and continuing for 12 months with taper at 9 months. Patients also receive methylprednisolone IV or orally beginning on day 8 and continuing for 7 months with taper at 4 months. Some patients may also receive methotrexate IV on days 1, 3 and 6.
  Interventions: Drug: busulfan; Drug: cyclophosphamide; Procedure: allogeneic bone marrow transplantation; Drug: methylprednisolone; Drug: methotrexate; Drug: cyclosporine

INTERVENTIONS:
Drug: busulfan — Given orally
  Other Names: BSF; BU; Misulfan; Mitosan; Myeloleukon; Myelosan
Drug: cyclophosphamide — Given IV
  Other Names: CPM; CTX; Cytoxan; Endoxan; Endoxana; Enduxan
Procedure: allogeneic bone marrow transplantation — Patients undergo allogeneic bone marrow transplant IV over 2-3 hours on day 0.
  Other Names: bone marrow therapy, allogeneic; bone marrow therapy, allogenic; transplantation, allogeneic bone marrow; transplantation, allogenic bone marrow
Drug: methylprednisolone — Given IV or orally
  Other Names: A-MethaPred; Depo-Medrol; Medrol; MePRDL; Solu-Medrol; Wyacort
Drug: methotrexate — Given IV
  Other Names: Abitrexate; amethopterin; Folex; methylaminopterin; Mexate; MTX
Drug: cyclosporine — Given IV or orally
  Other Names: 27-400; ciclosporin; cyclosporin; cyclosporin A; CYSP; Sandimmune

SUMMARY:
RATIONALE: Giving high doses of chemotherapy drugs, such as busulfan and cyclophosphamide, before a donor bone marrow transplant helps stop the growth of cancer cells. It may also stop the patient's immune system from rejecting the donor's stem cells. When the healthy stem cells from a donor are infused into the patient they may help the patient's bone marrow make stem cells, red blood cells, white blood cells, and platelets. Sometimes the transplanted cells from a donor can make an immune response against the body's normal cells. Giving cyclosporine, methylprednisolone, and methotrexate after transplant may stop this from happening.

PURPOSE: This clinical trial studies high-dose busulfan and high-dose cyclophosphamide followed by donor bone marrow transplant in treating patients with leukemia, myelodysplastic syndrome, multiple myeloma, or recurrent Hodgkin or Non-Hodgkin lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

I. To determine the toxicity and efficacy of the high-dose chemotherapy regimen which employs busulfan, cyclophosphamide, and allogeneic bone marrow transplantation.

II. To ascertain feasibility (safety) and efficacy of the use of intensive chemotherapy regimen (busulfan and cyclophosphamide) followed by allogeneic bone marrow transplantation in patients with leukemia, myelodysplastic syndromes, multiple myeloma, and lymphoma.

OUTLINE:

HIGH-DOSE CHEMOTHERAPY: Patients receive oral busulfan every 6 hours on days -8 to -5 and cyclophosphamide IV over 2 hours on days -4 and -3, or -4 to -2 .

TRANSPLANTATION: Patients undergo allogeneic bone marrow transplant IV over 2-3 hours on day 0.

GRAFT-VERSUS-HOST DISEASE PROPHYLAXIS: Patients receive cyclosporine IV over 6 hours on day -1, over 10 hours twice daily on days 0-20, and then orally every 12 hours beginning on day 21 and continuing for 12 months with taper at 9 months. Patients also receive methylprednisolone IV or orally beginning on day 8 and continuing for 7 months with taper at 4 months. Some patients may also receive methotrexate IV on days 1, 3 and 6 .

After completion of study treatment, patients are followed up periodically.

ELIGIBILITY:
Criteria

* Acute non-lymphocytic leukemia (FAB types M1-M7) in first, or second remission, or early first or second bone or marrow relapse (>31% marrow blasts and no circulating peripheral blasts)
* All patients with acute promyelocytic leukemia in first complete remission who have received retinoic acid and chemotherapy are not eligible
* Acute lymphocytic leukemia in first or second remission, or early first or second bone marrow relapse (31% marrow blasts and no circulating peripheral blasts)
* Pediatric ALL patients in first complete remission are not eligible
* Chronic myelogenous leukemia in first or second chronic phase, or accelerated phase
* Myelodysplastic syndrome =< 50 years
* Lymphoma patients age =< 50 years (non Hodgkins or Hodgkins) in first or second relapse, or refractory disease, who are ineligible for autologous bone marrow transplantation because of tumor in the bone marrow
* Multiple myeloma patients age =< 50 who have relapsed or are refractory to at least 2 chemo-radiation or chemotherapy regimens
* Patients who have failed a previous allogeneic bone marrow transplant
* Patients with inborn errors of metabolism
* ECOG performance status of 0 or 1
* Karnofsky performance status of >= 70%
* Patients must be HTLV-III (HIV) anti-body negative
* Acute and chronic leukemia patients must be age =< 50 years; patients up to age 60 years for any of these diseases who have a syngeneic donor are eligible
* Patients (or bone marrow donors) who are HTLV-III (HIV) antibody positive are ineligible for this study
* Patients must not have active infection
* Patients must not have cytotoxic chemotherapeutic agents for at least 4 weeks before the transplant conditioning regimen is to begin
* It is recommended but not required that acute leukemia patients undergoing transplantation in first remission must have received at least one course of consolidation therapy
* Patients undergoing transplant in early relapse are eligible for transplant in first and second relapse only
* Patients must have no history of acute myocardial infarction in the 6 months prior to transplantation, angina pectoris requiring nitrate therapy, uncontrolled major ventricular dysrhythmia, uncontrolled hypertension, or uncontrolled congestive heart failure
* A gated-pool radionuclide scan fraction must be >= 50%
* Serum creatinine must be =< 1.8% and a 24 hour creatinine clearance must be >= 60ml/min
* Serum direct bilirubin >= 1.8mg%, or serum SGOT or SGPT > twice normal will exclude patients from this study
* Severe symptomatic CNS disease of any etiology other than CNS leukemia will exclude patients from study
* FEV1 and DLco (corrected) must be >= 60% of normal
* pO2 > 60mmHg
* Insulin-dependent diabetes mellitus or uncompensated major thyroid or adrenal dysfunction render patients ineligible
* Written informed consent must be obtained
* Patients treated previously with radiation therapy in excess of 1000 cGy (rads) to any thoracic or abdominal port, or in excess of 3000 cGy (rads) to cranial-spinal ports, who are not eligible for other protocols are eligible for this study
* DONOR: All genotypically HLA- or D/DR identical siblings are eligible to be bone marrow donors so long as their general medical condition permits the safe use of general or spinal anesthesia; selected donors who are not HLA-identical may be considered for use as long as they are D/DR identical, MLC compatible, and are in good condition to safely undergo spinal or general anesthesia
* DONOR: This protocol will allow the use of donors who are unrelated but are HLA-A, b, C, D/Dr identical and MLC (mixed lymphocyte culture) compatible
* Patient must have adequate insurance to cover the cost of the transplant and hospitalization

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 1988-03; Primary Completion 2000-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Response rate | obtained at least one month apart beginning no earlier than two month after marrow infusion
  no evidence of leukemia as judged by two peripheral blood smears and two bone marrow aspirates and biopsies. Disease-free and overall survival data will be computed from the day of marrow infusion.
Toxicity as assessed by NCI CTC and engraftment (bone marrow) toxicity criteria | twice weekly

CONTACTS AND LOCATIONS:
Overall Officials: Hillard Lazarus, Principal Investigator — Ireland Cancer Center at University Hospitals Case Medical Center, Case Comprehensive Cancer Center
Locations (1):
- Ireland Cancer Center at University Hospitals Case Medical Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States